CLINICAL TRIAL: NCT00004311
Title: Phase II Study of the Effect of Leuprolide Acetate and Spironolactone on Insulin Resistance in Hyperandrogenic Women With Polycystic Ovarian Disease or Hyperandrogenism Insulin Resistance Acanthosis Nigricans Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Baylor College of Medicine (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11816; BCM-467
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-05

CONDITIONS: Acanthosis Nigricans; Polycystic Ovary Syndrome
Keywords: acanthosis nigricans; dermatologic disorders; endocrine disorders; polycystic ovarian syndrome; rare disease
MeSH Terms: conditions — Acanthosis Nigricans; Polycystic Ovary Syndrome; Skin Diseases; Endocrine System Diseases; Rare Diseases | interventions — Leuprolide; Spironolactone

INTERVENTIONS:
Drug: leuprolide acetate
Drug: spironolactone

SUMMARY:
OBJECTIVES: I. Evaluate insulin resistance in thin and obese hyperandrogenic women with polycystic ovarian disease or hyperandrogenism insulin resistance acanthosis nigricans syndrome and in thin and obese controls, using an estimation of tissue sensitivity to insulin.

II. Evaluate the effect of androgen suppression with leuprolide acetate and spironolactone on insulin secretion and resistance.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Participants are treated with subcutaneous leuprolide acetate followed by oral spironolactone. Each treatment is administered daily for 6 weeks, with a 6-week washout between drugs.

Patients and controls are alternately assigned to begin treatment with leuprolide acetate or spironolactone.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Polycystic ovarian disease Oligomenorrhea or amenorrhea Hirsutism Hyperandrogenism Hyperandrogenism insulin resistance acanthosis nigricans syndrome Hyperandrogenism Oligomenorrhea or amenorrhea Insulin resistance Acanthosis nigricans Hematocrit at least 30% Women with normal menstrual cycles not using oral contraception entered as controls

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-07; Study Completion 1996-01

CONTACTS AND LOCATIONS:
Overall Officials: Karen E. Elkind-Hirsch, Study Chair — Baylor College of Medicine